CLINICAL TRIAL: NCT01086332
Title: A Phase I/II Trial of the HIV Protease Inhibitor Nelfinavir and Concurrent Radiation and Chemotherapy in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Evaluation of Nelfinavir and Chemoradiation for Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Toxicities, lack of funding
Sponsor: University of Iowa (Other)
Collaborators: Holden Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Bryan Allen, Assistant Professor of Radiation Oncology, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200905705
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Pancreatic Neoplasms
Keywords: radiotherapy; gemcitabine; nelfinavir; neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Nelfinavir; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- phase 1/2 (Experimental): An escalating study of gemcitabine when combined with 1250 mg of nelfinavir twice daily. Dose of gemcitabine is increased for new subjects based on the experiences and tolerance of prior subjects. When the maximum tolerated dose is identified, a recommended phase 2 dose will be assigned and further subjects will receive that dose.
  Interventions: Drug: Nelfinavir; Drug: Gemcitabine

INTERVENTIONS:
Drug: Nelfinavir — 1250 mg twice daily
  Other Names: Viracept
Drug: Gemcitabine — Escalating doses of gemcitabine during concurrent radiation and nelfinavir therapy.
  Other Names: Gemzar

SUMMARY:
This study is designed to evaluate if nelfinavir works as a radiation sensitizer in combination with gemcitabine (a chemotherapy). We are also looking to establish the maximum dose of gemcitabine that is tolerated with the nelfinavir and radiation therapy, so the dose of gemcitabine is increased based on how previous trial participants tolerated their dose of gemcitabine.

DETAILED DESCRIPTION:
This trial utilizes gemcitabine (a chemotherapy agent commonly used for pancreatic cancer) and nelfinavir (an anti-retroviral agent FDA-approved for use in HIV+ patients) in addition to radiation therapy for treatment of borderline resectable pancreatic cancer. The trial seeks to determine the maximum tolerated dose of gemcitabine when administered concurrently with radiation therapy and 1250 mg nelfinavir twice daily.

The gemcitabine and radiation is standard; the dose of gemcitabine does vary nationally and internationally as to what the 'best dose' is. Administered weekly, doses can range from 400 mg/m2 to 1000 mg/m2. Thus, this is why the proposed clinical trial escalates the gemcitabine.

The gemcitabine will be administered weekly during radiation therapy for a total of 6 cycles. After completion of radiation therapy, the subjects will be evaluated by the surgeons for resectability. This ends the active portion of the clinical trial; the subjects will be followed for long-term progression free survival and for overall survival.

Primary endpoints for this trial are identifying the maximum tolerated dose of gemcitabine when administered concurrently with nelfinavir and radiation therapy (the phase I portion of this study) and the rate of resectability (typically, utilizing gemcitabine plus radiation therapy will convert up to 30% of patients from borderline resectable to resectable) for the phase II portion of the study.

Interim analyses and stopping rules are in place if an effect size is not observed in the therapeutic group compared to published reports of response to standard chemoradiation for borderline resectable cases.

ELIGIBILITY:
Closed to accrual.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities | Six weeks
  Evaluating adverse events and their association to the treatment to determine the recommended phase II dose of gemcitabine.

SECONDARY OUTCOMES:
Surgical resection rate | 8 weeks
  Evaluate the number of subjects who are now surgically resectable and then correlate the pathological outcomes with treatment (i.e., tumor cell kill).

CONTACTS AND LOCATIONS:
Overall Officials: Bryan G. Allen, M.D., PhD, Study Director — University of Iowa

IPD SHARING:
Plan to Share IPD: Yes
Data are shared upon request. Contact the clinical research team.
Supporting Information: Study Protocol, ICF
Time Frame: Upon request
Access Criteria: Depending upon the data desired, a confidentiality / non-disclosure agreement may be required.

REFERENCES:
- [Background] Plastaras JP, Vapiwala N, Ahmed MS, Gudonis D, Cerniglia GJ, Feldman MD, Frank I, Gupta AK. Validation and toxicity of PI3K/Akt pathway inhibition by HIV protease inhibitors in humans. Cancer Biol Ther. 2008 May;7(5):628-35. doi: 10.4161/cbt.7.5.5728. Epub 2008 May 14. PMID 18285707
- [Background] Gupta AK, Li B, Cerniglia GJ, Ahmed MS, Hahn SM, Maity A. The HIV protease inhibitor nelfinavir downregulates Akt phosphorylation by inhibiting proteasomal activity and inducing the unfolded protein response. Neoplasia. 2007 Apr;9(4):271-8. doi: 10.1593/neo.07124. PMID 17460771
- [Background] Pore N, Gupta AK, Cerniglia GJ, Jiang Z, Bernhard EJ, Evans SM, Koch CJ, Hahn SM, Maity A. Nelfinavir down-regulates hypoxia-inducible factor 1alpha and VEGF expression and increases tumor oxygenation: implications for radiotherapy. Cancer Res. 2006 Sep 15;66(18):9252-9. doi: 10.1158/0008-5472.CAN-06-1239. PMID 16982770
- [Background] Gupta AK, Cerniglia GJ, Mick R, McKenna WG, Muschel RJ. HIV protease inhibitors block Akt signaling and radiosensitize tumor cells both in vitro and in vivo. Cancer Res. 2005 Sep 15;65(18):8256-65. doi: 10.1158/0008-5472.CAN-05-1220. PMID 16166302